CLINICAL TRIAL: NCT05132101
Title: Analysis of the Real-world Prescription Pattern of Palbociclib Combination Therapy With Aromatase Inhibitor as a 1st Line Therapy in Metastatic Breast Cancer Patients Using the National Health Insurance Claims Data in South Korea
Brief Title: Analysis of the Real-world Prescription Pattern of Palbociclib Combination Therapy With Aromatase Inhibitor as a First Line Therapy in Metastatic Breast Cancer Patients Using the National Health Insurance Claims Data in South Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481167; Palbociclib HIRA (Other: Alias Study Number)
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Hormone receptor positive (HR+); Human Epidermal Growth Factor Receptor 2 Negative (HER2-); Metastatic Breast Cancer (MBC)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Patients who received Palbociclib as first line therapy in MBC setting — Patients who received Palbociclib as first line therapy in MBC setting

SUMMARY:
The objective of this study is to evaluate the real-world prescription patterns of Palbociclib in breast cancer (BC) patients who were treated with Palbociclib in combination with AI as a 1st line of therapy using the national health insurance claims data in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were prescribed with palbociclib in combination with AI for at least 1 cycle during the index period
* Patients who were diagnosed with BC during the index period

Exclusion Criteria:

* Male
* Prescribed with palbociclib during 12-month period preceding the index date

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: BC patients who were prescribed with Palbociclib in combination with AI for at least 1 cycle during the index period will be selected as the study population.
Sampling Method: Probability Sample
Enrollment: 2758 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Total treatment duration and cycle for Palbociclib | From index date (Index date: 06 Nov 2012 to 30 Sep 2020) to the end date of last palbociclib prescription (maximum of 34.8 months from the index date)

SECONDARY OUTCOMES:
Assessment on dose modification of Palbociclib as first line of therapy in BC patients in real-world setting. | From the index date (Index date: 06 Nov 2012 to 30 Sep 2020) to the time of reduction or increase in the dose given in the subsequent Palbociclib prescription (up to 30 Sep 2020)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Local Country Office, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481167